CLINICAL TRIAL: NCT06730126
Title: A Phase 2a Study of the ITK Inhibitor Soquelitinib to Reduce Lymphoproliferation and Improve Cytopenias in Autoimmune Lymphoproliferative Syndrome (ALPS)-FAS Patients
Brief Title: Study of the ITK Inhibitor Soquelitinib to Reduce Lymphoproliferation and Improve Cytopenias in Autoimmune Lymphoproliferative Syndrome (ALPS)-FAS Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001824; 001824-I
Record Dates: First submitted 2024-12-11; First posted 2024-12-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-11-28

CONDITIONS: Autoimmune Lymphoproliferative Syndrome
Keywords: Autoimmune Lymphoproliferative Syndrome; Fas; Hypersplenism; Lymphoproliferation; Interleukin-2 Inducible T-cell Kinase; Soquelitinib; Targeted Treatment
MeSH Terms: conditions — Autoimmune Lymphoproliferative Syndrome; Autoimmune Lymphoproliferative Syndrome, Type IA; Hypersplenism

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): The initial dosage for stage 1 of this study is 200 mg twice daily for up to 360 days. If stage 1 is repeated because there are no successes at this dosage, then it will be increased to 400 mg twice daily for up to 360 days. Alternatively, if there are safety concerns at either dosage, then it will be decreased to 100 mg twice daily for up to 360 days.
  Interventions: Drug: Soquelitinib

INTERVENTIONS:
Drug: Soquelitinib — Soquelitinib is an ITK inhibitor in clinical development for treating relapsed/refractory T-cell lymphoma.

SUMMARY:
Background:

Autoimmune lymphoproliferative syndrome (ALPS) is a rare disorder of the immune system caused by a mutation in the FAS gene. In ALPS, the body stores too many germ-fighting cells called lymphocytes. This can lead to an enlarged spleen and lymph nodes. Current treatments for ALPS can have many adverse effects. Better treatments for ALPS are needed.

Objective:

To test a study drug (soquelitinib) in people with ALPS.

Eligibility:

People aged 16 years and older with ALPS.

Design:

Participants will have 8 clinic visits and 6 remote visits within 1 year.

Participants will be screened. They will have a physical exam with blood and urine tests. Some may have tests of their lung function.

Soquelitinib is a tablet taken by mouth twice a day. Participants will record their doses and any symptoms on a paper or online form.

Blood tests and other procedures will be repeated during study visits. Three visits will include imaging scans. Participants will lie on a table that slides through a doughnut-shaped machine while X-rays capture pictures of the inside of their body.

Some participants may be able to remain in the study for a second year.

DETAILED DESCRIPTION:
Study Description:

This is a multisite open-label phase 2a study to evaluate the safety, tolerability, and preliminary efficacy of the interleukin (IL)-2 inducible Tcell kinase (ITK) inhibitor soquelitinib for treating ALPS-FAS. This study will be conducted in two stages, though the first stage may be repeated. In the first stage, 8 participants will be enrolled to receive 200 mg of soquelitinib twice daily for up to 360 days, with approximately monthly study visits (in person or remote). A safety and futility interim analysis will be conducted after all 8 participants have had a computed tomography (CT) or positron emission tomography (PET)/CT scan at day 90 and have completed at least 80% of their study drug regimen. If at least one participant has a positive response to the study drug and there are no safety concerns among the 8 participants, then the study will proceed to stage 2, in which 6 new participants will be enrolled and receive the same dosage as stage 1 (200 mg twice daily for 360 days).

If no stage 1 participant demonstrates a positive response to study drug but there are no safety concerns, then stage 1 will be repeated at a dosage of 400 mg twice daily for up to 360 days. New participants may be enrolled and/or the previous stage 1 participants may continue following a 90-day study drug washout. The safety and futility interim analysis will be repeated after all 8 participants have had a CT or PET/CT scan at day 90 and have completed at least 80% of their study drug regimen. Again, if there is at least 1 positive response and no safety concerns among these 8 participants, then the study will proceed to stage 2, in which 6 new participants will be enrolled and receive soquelitinib at 400 mg twice daily for up to 360 days.

The primary endpoints will be assessed after all 6 participants of stage 2 have had a CT or PET/CT scan at day 90 and have completed at least 80% of their study drug regimen. The trial will automatically be determined a failure if safety concerns or lack of positive response prevent procession to stage 2.

Primary Objectives:

To determine the efficacy of soquelitinib in reducing spleen volume or target lymph node volume in people with ALPS-FAS.

Secondary Objective:

1. To determine the efficacy of soquelitinib in improvement of lymphoproliferation and autoimmune disease, including cytopenias, in

   people with ALPS-FAS.
2. To determine the safety and tolerability of soquelitinib in people with ALPS-FAS.

Primary Endpoints:

Reduction of spleen volume or target lymph node volume by 25% from baseline to day 90, assessed by CT or PET/CT scan.

Secondary Endpoints:

1. Shrinkage in spleen volume from baseline to day 90.
2. Shrinkage in target lymph node volume from baseline to day 90.
3. Reduction of cytopenias by one severity level from baseline to day 90.
4. Reduction in prednisone dosage.
5. Grade 3 or 4 systemic infections within 360 days.
6. Clinically significant worsening of viral, mycobacterial, or fungal infection requiring new treatment or change of treatment by day 360.
7. Any drug-related grade 3 or 4 adverse event (AE) that triggers a pause.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Aged >= 16 years.
2. Able to provide informed consent (for ages >= 18 years) or has a parent(s) or guardian(s) who can provide permission to participate on their behalf (for ages <18 years).
3. Has a documented diagnosis of ALPS-FAS.
4. Has clinical evidence of active disease, defined as at least one enlarged lymph node and/or enlarged spleen.
5. If currently on corticosteroid therapy, then dose is less than 20 mg/day (prednisone equivalent) and has been stable for at least 4 weeks.
6. For participants to be seen at the NIH CC, co-enrolled on NIH protocol 93-I-0063.
7. Participants who can become pregnant or who can impregnate their partner must agree to either remain sexually abstinent or use two highly effective methods of contraception when engaging in sexual activities that can result in pregnancy, beginning 28 days before baseline until 3 months after the last dose. One method must be a barrier (eg, internal or external condom, cervical cap, or diaphragm). The second method may be any of the following:

7a. Oral contraceptive pill or hormonal patch or ring.

7b. Parenteral hormonal contraceptive implant.

7c. Intrauterine device.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Profound grade 3 or 4 cytopenias that cannot be improved with immunomodulatory treatments prior to enrolling in the clinical trial and starting the study drug. Per investigator discretion, individuals on a single agent may be included if the dose is stable for 12 weeks at screening and is not expected to confer additive toxicity.
2. Renal impairment, defined as serum creatinine >1.5 mg/dL (or 133 micromol/L) or estimated glomerular filtration rate <60 mL/min/1.73 m^2.
3. Liver impairment, defined as bilirubin, alanine aminotransferase, or aspartate aminotransferase greater than 2.5 times the upper limit of normal.
4. History of EBV-associated lymphoma.
5. Active EBV infection with EBV load >300 copies/mL.
6. Tuberculosis infection (active or latent) or undergoing tuberculosis treatment.
7. Infection with HIV or hepatitis B or C.
8. Current other invasive or systemic fungal, bacterial, or viral infection requiring therapy.
9. History of opportunistic infection within the previous 180 days.
10. History of invasive malignancy that required systemic therapy within the last 3 years.
11. Current use of moderate or strong cytochrome P450 isozyme (CYP)3A inhibitors or inducers that cannot be stopped before day 0.
12. Current use of P-glycoprotein (P-gp) inhibitors that cannot be stopped before day 0.
13. Known hypersensitivity or contraindication to CT contrast agent.
14. Pregnant or breastfeeding.
15. Any condition that, in the opinion of the study team contraindicates participation in this study.

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of spleen volume or target lymph node volume by 25% from baseline to day 90, assessed by CT or PET/CT scan. | Day 90
  To determine the efficacy of soquelitinib in reducing spleen volume or target lymph node volume in people with ALPS-FAS.

SECONDARY OUTCOMES:
Shrinkage in spleen volume from baseline to day 90. | Day 90
  To determine the efficacy of soquelitinib in improvement in lymphoproliferation and autoimmune disease, including cytopenias, in people with ALPS-FAS.
Shrinkage in target lymph node volume from baseline to day 90. | Day 90
  To determine the efficacy of soquelitinib in improvement in lymphoproliferation and autoimmune disease, including cytopenias, in people with ALPS-FAS.
Reduction of cytopenias by one severity level from baseline to day 90 | Day 90
  To determine the efficacy of soquelitinib in improvement in lymphoproliferation and autoimmune disease, including cytopenias, in people with ALPS-FAS and to determine the safety and tolerability of soquelitinib in people with ALPS-FAS.
Reduction in prednisone dosage. | End of Study
  To determine the efficacy of soquelitinib in improvement in lymphoproliferation and autoimmune disease, including cytopenias, in people with ALPS-FAS
Grade 3 or 4 systemic infections within 360 days. | Day 360
  To determine the safety and tolerability of soquelitinib in people with ALPS-FAS.
Clinically significant worsening of viral, mycobacterial, or fungal infection requiring new treatment or change of treatment by day 360. | End of Study
  To determine the safety and tolerability of soquelitinib in people with ALPS-FAS.
Any drug-related grade 3 or 4 AE AE that triggers a pause. | End of Study
  To determine the safety and tolerability of soquelitinib in people with ALPS-FAS.

CONTACTS AND LOCATIONS:
Overall Officials: V. Koneti Rao, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Clinical, laboratory, imaging and demographic data.
Supporting Information: Study Protocol, ICF
Time Frame: Following interim review and/or completion of study.
Access Criteria: Requests are reviewed by PI.

REFERENCES:
- [Background] Price S, Shaw PA, Seitz A, Joshi G, Davis J, Niemela JE, Perkins K, Hornung RL, Folio L, Rosenberg PS, Puck JM, Hsu AP, Lo B, Pittaluga S, Jaffe ES, Fleisher TA, Rao VK, Lenardo MJ. Natural history of autoimmune lymphoproliferative syndrome associated with FAS gene mutations. Blood. 2014 Mar 27;123(13):1989-99. doi: 10.1182/blood-2013-10-535393. Epub 2014 Jan 7. PMID 24398331
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001824-I.html